CLINICAL TRIAL: NCT03118492
Title: A Pilot Study of Reduced Intensity HLA-Haploidentical Hematopoietic Cell Transplantation With Post-Transplant Cyclophosphamide in Patients With Advanced Myelofibrosis
Brief Title: Combination Chemotherapy, Total Body Irradiation, and Donor Blood Stem Cell Transplant in Treating Patients With Secondary Myelofibrosis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16420; NCI-2017-00613 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16420 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Secondary Myelofibrosis
MeSH Terms: interventions — Stem Cell Transplantation; Cyclophosphamide; fludarabine; Melphalan; Mycophenolic Acid; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (combination chemotherapy, TBI, HCT) (Experimental): Patients receive melphalan IV over 30 minutes on day -5, fludarabine IV over 30-60 minutes on days -5 to -2. Patients undergo TBI on day -1 and HCT on day 0. Patients receive cyclophosphamide IV over 1-2 hours on days 3 and 4. Starting on day 5, patients receive tacrolimus IV then PO for 6 months followed by a taper, mycophenolate mofetil PO TID until day 35, and G-CSF IV daily until absolute neutrophil count > 1,500/mm^3 for 3 consecutive days. Treatment continues in the absence of disease progression or unexpected toxicity.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Glycosylated Recombinant Human G-CSF AVI-014; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Biological: Glycosylated Recombinant Human G-CSF AVI-014 — Given IV
  Other Names: AVI-014
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mycophenolate Mofetil — Given PO
  Other Names: CellCept; MMF
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TBI; Total Body Irradiation; Whole Body Irradiation; Whole-Body Irradiation

SUMMARY:
This pilot phase I trial studies the side effects of combination chemotherapy, total body irradiation, and donor blood stem cell transplant in treating patients with secondary myelofibrosis. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill cancer cells and shrink tumors. Giving combination chemotherapy and total body irradiation before a donor blood stem cell transplant helps to stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of reduced-intensity (fludarabine/melphalan) haploidentical hematopoietic cell transplantation (Haplo-HCT) followed by post-transplant cyclophosphamide (PTCy) in patients with advanced myelofibrosis (MF), as assessed by the evaluation of toxicities, including type, frequency, severity, attribution, time course and duration.

SECONDARY OBJECTIVES:

I. To summarize and evaluate hematologic (neutrophil and platelet) recovery. II. To evaluate and describe cytokine release syndrome (CRS) post haploidentical HCT in the setting of advanced myelofibrosis, as assessed by grade, frequency, severity, duration and reversibility (outcome).

III. To estimate graft failure-free survival (GFS) at 100-days post-transplant. IV. To estimate overall survival (OS), progression-free survival (PFS) and cumulative incidence (CI) of relapse/progression, and non-relapse mortality (NRM) at 100-days, 1-year, and 2-year post transplant.

V. To estimate the cumulative incidence of acute graft-versus-host disease (GvHD), grade II-IV, at 100-days post-transplant (per Keystone Consensus modification of the Glucksberg criteria).

VI. To estimate the cumulative incidence of chronic GvHD at 1-year and 2-year post transplant (per National Institutes of Health [NIH] Consensus Criteria).

VII. To characterize the severity and extent of acute and chronic GvHD.

EXPLORATORY OBJECTIVE:

I. To conduct correlative studies and describe inflammatory cytokine levels and GVHD biomarker levels in plasma and T cell differentiation/functions in patients enrolled onto the trial.

OUTLINE:

Patients receive melphalan intravenously (IV) over 30 minutes on day -5, fludarabine IV over 30-60 minutes on days -5 to -2. Patients undergo total body irradiation (TBI) on day -1 and hematopoietic cell transplantation (HCT) on day 0. Patients receive cyclophosphamide IV over 1-2 hours on days 3 and 4. Starting on day 5, patients receive tacrolimus IV then orally (PO) for 6 months followed by a taper, mycophenolate mofetil PO thrice daily (TID) until day 35, and glycosylated recombinant human G-CSF AVI-014 (G-CSF) IV daily until absolute neutrophil count > 1,500/mm^3 for 3 consecutive days. Treatment continues in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are followed for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary of secondary myelofibrosis with transplant indication by Dynamic International Prognostic Scoring System (DIPSS)-plus (> intermediate-1)
* Patients >= age 50 must have a comorbidity score (hematopoietic cell transplant-comorbidity index [HCT-CI]) < 4 (Sorror)
* Patients can be in chronic phase (CP) with bone marrow (BM) blast count =< 15% as long as no evidence of disease acceleration per principal investigator (PI) and treating physician's opinion or after progression to acute myeloid leukemia (AML) and achieved =< 5% BM blasts (morphologic complete remission [CR] prior to transplant)
* Lack of an human leukocyte antigen (HLA) matched donor or need to proceed fast to transplantation when a patient does not have an immediately available matched unrelated donor (typed by high-resolution in the registry)
* Performance status >= 70% (Karnofsky); patients > 50 years should have adequate cognitive function; any concerns regarding cognitive function should be addressed by a geriatrician/neurologist
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST)/bilirubin =< 5 X upper limit of normal (ULN)
* Measured creatinine clearance > 60 mls/min
* Left ventricular ejection fraction (LVEF) >= 50%
* Corrected carbon monoxide diffusing capability (DLCOc) >= 50%
* No active infections
* Prior treatment with JAK2 inhibitor therapy is not excluded; a JAK2 inhibitor will need to be stopped 1-2 days prior to starting conditioning regimen
* DONOR: Documented informed consent per local, state and federal guidelines
* DONOR: Genotypically haploidentical as determined by HLA typing

  * Preferably a non-maternal HLA haploidentical relative due to data of high incidence of graft failure with use of maternal HLA haploidentical cells
  * Eligible donors include biological parents, siblings or half-siblings, children, or cousins in rare instances
* DONOR: Absence of pre-existing donor-specific anti-HLA antibodies (DSA) in the recipient; Patients with pre-existing DSA could undergo desensitization per City of Hope (COH) standard operating procedures [SOP] and should have DSA < MFI of 2000 prior to conditioning at discretion of PI
* DONOR: Infectious disease screening performed within 30 days prior to stem cell mobilization per federal guidelines and is:

  * Seronegative for HIV 1+2 antibody (Ab) and/or HIV polymerase chain reaction (PCR), human T-cell leukemia virus (HTLV) I/II Ab, hepatitis B virus surface antigen (HBsAg), hepatitis B virus surface antibody (HBcAb), hepatitis C virus (HCV) Ab
  * Negative rapid plasma reagin (RPR) for syphilis
* DONOR: Women of childbearing potential (WOCBP): Urine pregnancy testing performed within 7 days prior to stem cell mobilization
* DONOR: Is approved and completed evaluation prior to recipient initiation of the preparative regimen per institutional guidelines

Exclusion Criteria:

* Evidence of severe portal hypertension with evidence of decompensation either with bleeding varices, large volume ascites, or hepatic encephalopathy
* In a bone marrow biopsy 4 weeks prior to start of conditioning on study:

  * > 15% bone marrow blasts at transplant if no history of AML and per PI and treating physician's opinion of disease acceleration
  * > 5% if had previous progression to AML
* Human immunodeficiency virus (HIV) positive; active hepatitis B or C
* Patients with active infections; the PI is the final arbiter of the eligibility
* Patients with evidence of severe pulmonary hypertension by echocardiogram and confirmed by a subsequent right side cardiac catheterization pre-enrollment
* Liver cirrhosis
* Prior central nervous system (CNS) involvement by tumor cells
* History of another primary malignancy that has not been in remission for at least 3 years (the following are exempt from the 3-year limit: non-melanoma skin cancer, fully excised melanoma in situ [stage 0], curatively treated localized prostate cancer, and cervical or breast carcinoma in situ on biopsy or a squamous intraepithelial lesion on papanicolaou [PAP] smear)
* Positive beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization
* Noncompliance - inability or unwillingness to comply with medical recommendations regarding therapy or follow-up, including smoking tobacco
* DONOR: Has undergone solid organ, stem cell, bone marrow or blood transplantation
* DONOR: Receiving any investigational agents, or concurrent biological, chemotherapy, immunosuppression or radiation therapy
* DONOR: Active infection
* DONOR: Thrombocytopenia < 150,000 cells /mm^3 at baseline evaluation
* DONOR: Sero-positive for HIV-1 & 2 antibody, HTLV-I & II antibody, hepatitis B virus (HBV) and HCV
* DONOR: Medical or physical reason which makes the donor unlikely to tolerate or cooperate with growth factor therapy and leukapheresis
* DONOR: Factors which place the donor at increased risk for complications from leukapheresis or G-CSF therapy
* DONOR: WOCBP: Pregnant or =< 6 months breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2026-05-26 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 100 days post-hematopoietic cell transplantation (HCT)
  Assessed by Bearman Toxicity Scale and National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version (CTCAE) 4.03. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study regimen and reversibility or outcome.
Incidence of unacceptable toxicity | Up to 2 years
  Assessed by Bearman Toxicity Scale and NCI CTCAE version 4.03. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study regimen and reversibility or outcome.

SECONDARY OUTCOMES:
Neutrophil recovery | Up to 2 years
  Defined as the first of 3 measurements on different days when the patient has an absolute neutrophil count of >= 500/uL after conditioning.
Platelet recovery | Up to 2 years
  Defined as the first day of a minimum of 3 measurements on different days that the patient has achieved a platelet count >= 20,000/uL and did not receive a platelet transfusion in the previous 7 days.
Incidence of cytokine release syndrome (CRS) | After haploidentical HCT, assessed up to 2 years
  Defined and graded per American Society for Transplantation and Cellular Therapy (ASTCT) criteria.
Graft failure-free survival | Time from start of protocol treatment/infusion of stem cell product to graft-failure, death (from any cause), or last contact, whichever occurs first, assessed up to 2 years
  Will be calculated using Kaplan-Meier product-limit method, 95% confidence intervals will be calculated.
Overall survival | Time from start of protocol treatment/infusion of stem cell product to death (from any cause), or last contact, whichever occurs first, assessed up to 36 months
  Will be calculated using Kaplan-Meier product-limit method, 95% confidence intervals will be calculated.
Progression-free survival | Time from start of protocol treatment/infusion of stem cell product to, relapse, progression, death (from any cause), or last contact, whichever occurs first, assessed up to 2 years
  Will be calculated using Kaplan-Meier product-limit method, 95% confidence intervals will be calculated.
Cumulative incidence of relapse/progression | Up to 2 years
  The cumulative incidence of relapse/progression will be estimated using the method described by Gooley et al. (1999).
Non-relapse mortality (NRM) | Up to 2 years
  The cumulative incidence of NRM will be estimated using the method described by Gooley et al. (1999).
Cumulative incidence of acute graft versus host disease (GvHD) | Up to day 100 post-HCT
  Assessed by Keystone Consensus criteria. Time to the first day of acute GvHD onset (of any grade) will be used to estimate the cumulative incidence.
Cumulative incidence of chronic graft versus host disease GvHD | Up to 2 years post-HCT
  Assessed by National Institutes of Health Consensus Criteria. Time to the first day of chronic GvHD onset (of any grade) will be used to estimate the cumulative incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Monzr M Al Malki, Principal Investigator — City of Hope Medical Cancer Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States